CLINICAL TRIAL: NCT00064142
Title: A Phase II Trial of Topical Halofuginone in Patients With HIV Related Kaposi's Sarcoma
Brief Title: Halofuginone Hydrobromide in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02925; AMC-036; CDR0000309055; U01CA070019 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: AIDS-related Kaposi Sarcoma; Recurrent Kaposi Sarcoma
MeSH Terms: conditions — AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — halofuginone

ARMS (2):
- Arm I (halofuginone hydrobromide) (Experimental): Patients apply topical halofuginone hydrobromide ointment to each of 6 lesions twice a day for 12 weeks.
  Interventions: Drug: halofuginone hydrobromide; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (placebo) (Placebo Comparator): Patients apply topical placebo ointment to each of 6 lesions twice a day for 12 weeks.
  Interventions: Other: placebo; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: halofuginone hydrobromide — Applied topically
  Other Names: halofuginone; halofuginone HBr; RU 19110; Tempostatin
  Arms: Arm I (halofuginone hydrobromide)
Other: placebo — Applied topically
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies how well halofuginone hydrobromide works in treating patients with human immunodeficiency virus (HIV)-related Kaposi's sarcoma. Halofuginone hydrobromide ointment may stop the growth of Kaposi's sarcoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tumor response rate of acquired immune deficiency syndrome (AIDS)-related Kaposi's sarcoma to topical halofuginone (halofuginone hydrobromide) versus vehicle control.

II. To evaluate the safety and tolerability of topical halofuginone and vehicle in patients with AIDS-related Kaposi's sarcoma.

SECONDARY OBJECTIVES:

I. To determine the ability of topical halofuginone to inhibit expression of matrix metallopeptidase 2 (MMP-2) and Collagen type I in AIDS-related Kaposi's sarcoma.

II. To explore the relationship between baseline cluster of differentiation (CD) 4 and CD8 counts, HIV viral load and human herpesvirus 8 (HHV-8) viral load and response to halofuginone.

III. To characterize the pharmacokinetics of halofuginone.

OUTLINE: Twelve treatable Kaposi's sarcoma lesions are selected on each patient, and these 12 lesions are randomized equally to 1 of 2 treatment arms (6 lesions receive study treatment and 6 lesions receive placebo); each patient serves as his/her own control.

ARM I: Patients apply topical halofuginone hydrobromide ointment to each of 6 lesions twice a day for 12 weeks.

ARM II: Patients apply topical placebo ointment to each of 6 lesions twice a day for 12 weeks.

Patients with stable or responding disease in either or both groups of treated lesions (halofuginone hydrobromide ointment or placebo ointment) may receive open-label treatment with topical halofuginone hydrobromide ointment to all 12 lesions for an additional 12 weeks as above in the absence of disease progression or unacceptable toxicity.

Patients are followed for at least 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Kaposi's sarcoma with at least 14 cutaneous lesions, 12 of which are measurable in two dimensions and can serve as marker lesions; each of the 14 lesions must measure a minimum of 0.5 cm in diameter, so that a 4 mm punch biopsy will be entirely composed of Kaposi's sarcoma
* Serologic documentation of HIV infection by any of the Food and Drug Administration (FDA) approved tests
* Karnofsky performance status >= 60%
* Hemoglobin >= 8 g/dl
* Absolute neutrophil count >= 750 cells/mm^3
* Platelet count >= 75,000/mm^3
* Creatinine < 1.5 times the upper limit of normal or creatinine clearance >= 60 mL/min
* Total bilirubin should be =< 1.5 x upper limit of normal (ULN); if, however, the elevated bilirubin is felt to be secondary to indinavir therapy, patients will be allowed to enroll on protocol if the total bilirubin is =< 3.5 mg/dl provided that the direct bilirubin is normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x the upper limit of normal
* Life expectancy >= 3 months
* Ability and willingness to give informed consent; patients who are younger than 18 years of age will require the consent of a parent or guardian.
* All women of childbearing potential must have a negative serum b human chorionic gonadotropin (HCG) within 72 hours prior to study entry and must practice adequate birth control to prevent pregnancy while receiving treatment and for three months after treatment is discontinued
* Patients must, in the opinion of the investigator, be capable of complying with the protocol
* Patients receiving antiretroviral therapy must be on a stable regimen for at least 12 weeks prior to study entry without showing evidence of ongoing Kaposi's sarcoma (KS) regression (ie, less than 25% decrease in the size, number or nodularity of KS lesions in the opinion of the investigator); patients may receive any FDA approved antiretroviral therapy or agents available through a treatment IND; concurrent treatment with highly active antiretroviral therapy should be strongly encouraged, in accordance with DHHS guidelines (http://www.aids-ed.org/pdfs/adult_2-4-02.pdf) but will not be required for participation

Exclusion Criteria:

* Concurrent, acute, active, untreated opportunistic infection other than oral thrush or genital herpes within 14 days of enrollment
* Known active visceral Kaposi's sarcoma or symptomatic Kaposi's sarcoma-related edema that interferes with function or requires cytotoxic therapy
* Concurrent neoplasia requiring cytotoxic therapy
* Acute treatment for an infection (other than oral thrush or genital herpes) or other serious medical illness within 14 days of study entry
* Anti-neoplastic treatment for Kaposi's sarcoma (including chemotherapy, radiation therapy, local therapy, biological therapy, or investigational therapy) within four weeks of study entry
* Previous local therapy of any KS-indicator lesion within 60 days unless the lesion has clearly progressed since treatment
* Corticosteroid treatment, other than replacement doses
* Use of investigational agents other than antiretroviral drugs available under expanded access or compassionate use protocols
* Pregnant or breast feeding females are excluded from participation in this study since the effects of halofuginone on an unborn or young child are unknown and may potentially be toxic

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-05; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 30 days
  McNemar's chi-square test will be used to compare vehicle control and halofuginone with respect to response rates.
Safety of topical halofuginone as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 30 days after completion of treatment
  McNemar's chi-square test will be used to compare the two treatments with respect to the incidence of specific adverse events.

SECONDARY OUTCOMES:
Change in MMP-2 and collagen type I levels | From baseline to 4 weeks
Change in MMP-2 and collagen type I levels | From baseline to 12 weeks
  Changes from baseline in MMP-2 and Collagen type I for halofuginone and vehicle control lesions will be compared using the Wilcoxon rank sum test.
Relationship of CD4, CD8, HIV viral load and HHV-8 viral load on response | Up to 30 days
  Logistic regression analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Krown, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (1):
- AIDS - Associated Malignancies Clinical Trials Consortium, Rockville, Maryland, United States

REFERENCES:
- [Derived] Young SK, Baird TD, Wek RC. Translation Regulation of the Glutamyl-prolyl-tRNA Synthetase Gene EPRS through Bypass of Upstream Open Reading Frames with Noncanonical Initiation Codons. J Biol Chem. 2016 May 13;291(20):10824-35. doi: 10.1074/jbc.M116.722256. Epub 2016 Mar 21. PMID 27002157